CLINICAL TRIAL: NCT04317768
Title: The Effectiveness of Oral Health Education Using Audio-visual Aids and Frequent Motivation on Oral Health Status, Treatment Needs and Barriers to Care Among Children at Social Homes in Jordan
Brief Title: Effect of Oral Health Education on Oral Health Status, Treatment Needs and Barriers to Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: JUST 293-2018
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries; Gingivitis
Keywords: Oral health status; Dental treatment needs; Barriers to dental care; Children at social homes
MeSH Terms: conditions — Dental Caries; Gingivitis

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional study on a randomly selected group of children from randomly selected social homes in Jordan. Children and/or the care giver (n=500) will answer a questionnaire in an interview about his/her demographics, oral health related habits, the child general health status, the child oral health related quality of life, barriers to getting dental care, treatment needs for those children.
  A thorough clinical examination will be done to these children by a mouth mirror and explorer at a suitable room in the social home. The investigators will record the baseline oral health status parameters (Caries, gingival health and presence of plaque).
  For the interventions; A representative sample (25%) will be divided to two subgroups; group one (Study) and group two (Control) which will be matched for age and gender.
Who Masked: Outcomes Assessor
Masking Description: The statistician is blinded to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): They will be educated and motivated by an intensive program consisting of verbal instructions, Power Point lectures, posters and live demonstrations about oral hygiene instructions and teaching the proper way to brush the teeth. These will be reinforced by the investigator at intervals of 1 week, 1 month, 3 months, 6 months and 1 year.
  Interventions: Behavioral: Basic oral health education and motivation; Behavioral: Intensive oral health education and motivation
- Control group (Other): They will receive verbal oral hygiene instructions using a model to demonstrate only once at the beginning of the study, no further motivation or educational seminars will be done.
  Interventions: Behavioral: Basic oral health education and motivation

INTERVENTIONS:
Behavioral: Basic oral health education and motivation — Subjects will receive verbal oral hygiene instructions using a model to demonstrate only once at the beginning of the study, no further motivation or educational seminars will be done.
Behavioral: Intensive oral health education and motivation — Subjects will be educated and motivated by an intensive program consisting of verbal instructions, PowerPoint lectures, posters and live demonstrations about oral hygiene instructions and teaching the proper way to brush the teeth. These will be reinforced by the investigator at intervals of 1 week, 1 month, 3 months, 6 months and 1 year.
  Arms: Study group

SUMMARY:
Jordanian children have very poor oral hygiene parameters, and this is reflected as very high caries prevalence and poor gingival health conditions. This study will focus on children at social homes in the community in order to establish a baseline reference about their oral health status, treatment needs, and barriers to dental care. Also, to report the efficacy of oral health education using audio-visual aids and frequent motivation on oral health status, treatment needs and barriers to care among children at social homes in Jordan.

DETAILED DESCRIPTION:
The oral health status (OHS) for children and adults is a reflection of the whole body general health status as well as the overall quality of life. Jordanian children have very poor oral hygiene parameters, and this is reflected as very high caries prevalence and poor gingival health conditions. Orphans and children who come from broken homes are suspected to have poorer oral health conditions from their peers in the public due to the different parameters that can affect their general health in whole and oral health in particular, and this could affect their quality of life. These parameters can be related to socioeconomic status, psychological and behavioral conditions, access to care and other factors. The role of tooth brushing in decreasing dental caries and enhancing the gingival health is well-established in the literature, and oral health education programs have proven to be effective in improving the oral health knowledge, attitude and behavior of children. These programs could be regarded as an effective measure to enhance the oral health status and establish good routines in childhood which is vital for optimum oral health and provision of lifelong protection against caries.

This study will focus on children at social homes in the community in order to establish a baseline reference about their oral health status, treatment needs, and barriers to dental care. Also, to report the efficacy of oral health education using audio-visual aids and frequent motivation on oral health status, treatment needs and barriers to care among children at social homes in Jordan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children living in social homes among age group specified

Exclusion Criteria:

* Children with poor behavior

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Measure of dental caries | 1 year
  Decayed, missing, filled teeth
Gingival health | 1 year
  Presence or absence of gingival inflammation
Oral hygiene | 1 year
  Presence or absence of dental plaque

CONTACTS AND LOCATIONS:
Overall Officials: Ola Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No